CLINICAL TRIAL: NCT02824939
Title: Comparison of Ultrasound Guided Quadratus Lumborum Block With Ultrasound Guided TAP Block for Postoperative Analgesia After Laparoscopic Nephrectomy: a Prospective Randomized Controlled Trial
Brief Title: Comparison of Quadratus Lumborum Block With TAP Block for Postoperative Analgesia After Laparoscopic Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Kritika Rathour, Junior Resident, Department of Anaesthesia and Intensive Care, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NK/2663/MS/3121-22
Record Dates: First submitted 2016-06-27; First posted 2016-07-07 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Transversus Abdominis Plane group (Experimental)
  Interventions: Other: Transversus Abdominis Plane (TAP) Block
- Quadratus Lumborum group (Experimental)
  Interventions: Other: Quadratus Lumborum (QL) Block
- Control group (No Intervention)

INTERVENTIONS:
Other: Transversus Abdominis Plane (TAP) Block — 0.5 ml/kg of 0.25 % Bupivacaine deposited in the transversus abdominis plane under ultrasound guidance postoperatively
  Arms: Transversus Abdominis Plane group
Other: Quadratus Lumborum (QL) Block — 0.5 ml/kg of 0.25 % Bupivacaine deposited in the anterolateral aspect of the quadratus lumborum muscle under ultrasound guidance postoperatively
  Arms: Quadratus Lumborum group

SUMMARY:
This is a randomised controlled trial which will compare the Quadratus Lumborum (QL) Block with the Transversus Abdominis Plane (TAP) Block in terms of analgesic efficacy, ease of performance and safety when administered postoperatively in patients who undergo laparoscopic nephrectomy.

To fulfill this purpose, three groups of patients each with 32 patients, will be formed. Patients in the Transversus Abdominis Plane (TAP) group and Quadratus Lumborum (QL) group will each receive the respective blocks with 0.4 ml/kg of 0.25% Bupivacaine, after completion of surgery. The third (Control group) will not receive any blocks. After shifting patients to recovery all three groups will be put into intravenous patient controlled analgesia (PCA) Morphine as rescue analgesic regimen as per a set protocol. Morphine consumption over the first postoperative 24 hours, ease of performance of individual blocks and associated adverse events, adverse events associated with opioid use, patient recovery and satisfaction will be noted.

ELIGIBILITY:
Inclusion Criteria:

* patients between 18-65 years of age,
* ASA class I or II,
* undergoing elective unilateral laparoscopic nephrectomy
* under general anaesthesia

Exclusion Criteria:

Patients with any of the following:

* refusal to participate in the study
* coagulopathy/ thrombocytopenia
* localised infection at the proposed site of injection
* inability to comprehend the scoring systems to be employed or use PCA due to physical or mental problems
* known allergy to the drugs to be used (local anesthetics, opioids)
* opioid tolerance/ dependence
* renal impairment
* hepatic impairment
* known cardio-respiratory impairment
* morbid obesity/ sleep apnoea

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-09; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Cumulative morphine consumption in 24 hours in milligrams | within the first 24 hours after surgery

SECONDARY OUTCOMES:
Pain scores at rest and on movement as measured by numeric rating scale (0 to 10) | within the first 24 hours after surgery
Time to first demand of rescue analgesic in hours | within the first 24 hours after surgery
Ease of performing the respective blocks (assessed by time required to perform the blocks in minutes and number of attempts required to perform the blocks) | while performing block
Incidence of block related complications | within the first 24 hours after surgery
Incidence of adverse effects related to opioid use (derrived from incidence of nausea and vomiting, sedation and respiratory depression) | within the first 24 hours after surgery
Patient satisfaction as measured by numeric rating scale (0 to 10) | 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alexander JI. Pain after laparoscopy. Br J Anaesth. 1997 Sep;79(3):369-78. doi: 10.1093/bja/79.3.369. No abstract available. PMID 9389858
- [Background] Bisgaard T, Klarskov B, Rosenberg J, Kehlet H. Characteristics and prediction of early pain after laparoscopic cholecystectomy. Pain. 2001 Feb 15;90(3):261-269. doi: 10.1016/S0304-3959(00)00406-1. PMID 11207398
- [Background] Sjovall S, Kokki M, Kokki H. Laparoscopic surgery: a narrative review of pharmacotherapy in pain management. Drugs. 2015 Nov;75(16):1867-89. doi: 10.1007/s40265-015-0482-y. PMID 26493289
- [Background] Gorevski E, Wead S, Tevar A, Succop P, Volek P, Martin-Boone J. Retrospective evaluation of donor pain and pain management after laprascopic nephrectomy. Transplant Proc. 2011 Sep;43(7):2487-91. doi: 10.1016/j.transproceed.2011.06.038. PMID 21911110
- [Background] Rozen WM, Tran TM, Ashton MW, Barrington MJ, Ivanusic JJ, Taylor GI. Refining the course of the thoracolumbar nerves: a new understanding of the innervation of the anterior abdominal wall. Clin Anat. 2008 May;21(4):325-33. doi: 10.1002/ca.20621. PMID 18428988
- [Background] Mathuram Thiyagarajan U, Bagul A, Nicholson ML. Pain management in laparoscopic donor nephrectomy: a review. Pain Res Treat. 2012;2012:201852. doi: 10.1155/2012/201852. Epub 2012 Oct 23. PMID 23150820
- [Background] McDonnell JG, O'Donnell BD, Farrell T, Gough N, Tuite D, Power C, Laffey JG. Transversus abdominis plane block: a cadaveric and radiological evaluation. Reg Anesth Pain Med. 2007 Sep-Oct;32(5):399-404. doi: 10.1016/j.rapm.2007.03.011. PMID 17961838
- [Background] Barrington MJ, Ivanusic JJ, Rozen WM, Hebbard P. Spread of injectate after ultrasound-guided subcostal transversus abdominis plane block: a cadaveric study. Anaesthesia. 2009 Jul;64(7):745-50. doi: 10.1111/j.1365-2044.2009.05933.x. PMID 19624629
- [Background] Tran TM, Ivanusic JJ, Hebbard P, Barrington MJ. Determination of spread of injectate after ultrasound-guided transversus abdominis plane block: a cadaveric study. Br J Anaesth. 2009 Jan;102(1):123-7. doi: 10.1093/bja/aen344. PMID 19059922
- [Background] Lee TH, Barrington MJ, Tran TM, Wong D, Hebbard PD. Comparison of extent of sensory block following posterior and subcostal approaches to ultrasound-guided transversus abdominis plane block. Anaesth Intensive Care. 2010 May;38(3):452-60. doi: 10.1177/0310057X1003800307. PMID 20514952
- [Result] De Oliveira GS Jr, Castro-Alves LJ, Nader A, Kendall MC, McCarthy RJ. Transversus abdominis plane block to ameliorate postoperative pain outcomes after laparoscopic surgery: a meta-analysis of randomized controlled trials. Anesth Analg. 2014 Feb;118(2):454-463. doi: 10.1213/ANE.0000000000000066. PMID 24445643
- [Result] Carney J, Finnerty O, Rauf J, Bergin D, Laffey JG, Mc Donnell JG. Studies on the spread of local anaesthetic solution in transversus abdominis plane blocks. Anaesthesia. 2011 Nov;66(11):1023-30. doi: 10.1111/j.1365-2044.2011.06855.x. Epub 2011 Aug 18. PMID 21851346
- [Result] Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Nov;32(11):812-8. doi: 10.1097/EJA.0000000000000299. PMID 26225500
- [Result] Hosgood SA, Thiyagarajan UM, Nicholson HF, Jeyapalan I, Nicholson ML. Randomized clinical trial of transversus abdominis plane block versus placebo control in live-donor nephrectomy. Transplantation. 2012 Sep 15;94(5):520-5. doi: 10.1097/TP.0b013e31825c1697. PMID 22902793
- [Result] Baeriswyl M, Kirkham KR, Kern C, Albrecht E. The Analgesic Efficacy of Ultrasound-Guided Transversus Abdominis Plane Block in Adult Patients: A Meta-Analysis. Anesth Analg. 2015 Dec;121(6):1640-54. doi: 10.1213/ANE.0000000000000967. PMID 26397443
- [Result] Visoiu M, Yakovleva N. Continuous postoperative analgesia via quadratus lumborum block - an alternative to transversus abdominis plane block. Paediatr Anaesth. 2013 Oct;23(10):959-61. doi: 10.1111/pan.12240. Epub 2013 Aug 9. PMID 23927552
- [Result] Kadam VR. Ultrasound-guided quadratus lumborum block as a postoperative analgesic technique for laparotomy. J Anaesthesiol Clin Pharmacol. 2013 Oct;29(4):550-2. doi: 10.4103/0970-9185.119148. PMID 24249997
- [Result] Carvalho R, Segura E, Loureiro MD, Assuncao JP. [Quadratus lumborum block in chronic pain after abdominal hernia repair: case report]. Rev Bras Anestesiol. 2017 Jan-Feb;67(1):107-109. doi: 10.1016/j.bjan.2014.08.001. Epub 2014 Dec 6. Portuguese. PMID 25487690
- [Result] Chakraborty A, Goswami J, Patro V. Ultrasound-guided continuous quadratus lumborum block for postoperative analgesia in a pediatric patient. A A Case Rep. 2015 Feb 1;4(3):34-6. doi: 10.1213/XAA.0000000000000090. PMID 25642956